CLINICAL TRIAL: NCT02647307
Title: A Phase I, Open Label, Parallel Group Study to Evaluate the Effect of Ethnicity on the Pharmacokinetics, Pharmacodynamics and Safety of a DS 1040b IV Infusion Administered to Healthy Male Subjects
Brief Title: Study of the Effects of Ethnicity on the Pharmacokinetics, Pharmacodynamics and Safety of DS-1040b
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DS1040-A-E108; 2015-003470-32 (EudraCT Number)
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2016-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DS-1040b (Experimental): Single 12-hour intravenous infusion of DS-1040b (20 mg).
  Interventions: Drug: DS-1040b

INTERVENTIONS:
Drug: DS-1040b — Single 12-hour intravenous infusion of DS-1040b (20 mg)

SUMMARY:
The proposed study is not hypothesis testing but is intended to explore the effects of different ethnic groups (Caucasian, Japanese, Chinese, and Korean) on the PK (pharmacokinetic), PD (pharmacodynamic), and safety of an IV infusion of DS 1040b.

Subjects entering the study will receive a single 12 hour infusion of DS-1040b and be followed up to assess the effects on ethnicity on blood levels of DS-1040b as well as safety & tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged ≥ 18 years to 60 years, inclusive.
* Caucasian, Japanese, Chinese and Korean must have both parents and all 4 grandparents of equivalent descent.
* Subjects with a body mass index (BMI) of ≥ 18 kg/m2 to 30 kg/m2, inclusive, and weighing ≥ 50 kg to 100 kg, inclusive. BMI is calculated as weight [kg]/(height [m])2.
* Subjects must be in good health as determined by medical history, physical examination and Screening investigations, and taking no regular medication.
* Willing to comply with all study restrictions, including the use of contraception, concomitant medication and dietary and lifestyle restrictions.
* Possessing sufficient intelligence to understand the nature of the study and any hazards of participating in it, and the ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study.
* Has given written consent to participate after reading the informed consent form (ICF), and after having the opportunity to discuss the study with the Investigator or delegate.
* Have given written consent to have his data entered into The Overvolunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG findings or laboratory values that could interfere with the objectives of the study or the safety of the subject.
* Presence or history of acute or chronic illness, including (but not limited to) liver (Gilbert's Syndrome is permitted) or kidney disease, hypertension, seizures, or any known impairment of endocrine, or other specific body organ dysfunction.
* Presence or history of severe adverse reaction to any medicine.
* Presence or history of malignant disease.
* Significant illness within 4 weeks before the dose of study medication.
* Dosed in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical trials during the study and for 3 months after receipt of study medication.
* Participation in another clinical study with DS-1040b.
* Blood pressure (BP) and heart rate (HR) in semi supine position at the Screening examination outside the ranges 90 mmHg to 140 mmHg systolic, 40 mmHg to 90 mmHg diastolic; HR 40 beats/min to 100 beats/min. A subject with vital signs values outside the reference range for the population being studied may be included at the Investigator's discretion if it is unlikely to introduce additional risk factors and will not interfere with study procedures.
* Abnormal ECG waveform morphology at Screening that would preclude accurate measurement of the uncorrected QT interval (QT) duration.
* QT interval for HR corrected using Fridericia's formula (QTcF) interval duration > 430 msec obtained as an average from the measurements on triplicate Screening ECGs.
* Use of any prescription medicine, over the counter (OTC) medications, herbal remedies (such as St John's Wort), or food known to be strong inhibitors or strong inducers of cytochrome (CYP) enzymes during the 30 days before the dose of study medication; use of any other prescription or OTC medicine (except as permitted), including dietary supplements or herbal remedies, during the 7 days before receiving study medication.
* Consumption of certain foods or beverages before the dose and throughout the study period
* Loss of more than 400 mL blood (or plasma), or donation of platelets or other blood components during the 3 months before the dose of study medication, or unwilling to abstain from doing so during the study and for 3 months after receipt of study medication.
* Abuse of drugs or alcohol in the past, or intake of more than 21 units of alcohol weekly.
* Moderate to heavy use of tobacco products or nicotine containing products (eg ≥ 5 cigarettes per day during the 3 months before the dose of study medication.
* Male subjects have to agree to use contraception (condom with spermicide) in addition to having their female partner (if of childbearing potential) use another form of contraception (eg, an intrauterine device, diaphragm with spermicide, oral contraceptive, injectables, or subdermal hormonal implant) from receiving study medication until 4 months following the dose administration. Also, male subjects must not donate sperm until at least 4 months following the last dose administration.
* Evidence of acute or chronic infectious disease at Screening, including: positive Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus (HCV) antibody, or Human Immunodeficiency Virus (HIV) antibody.
* Subjects who have used anticoagulants (ie, warfarin, low molecular weight heparin, thrombin inhibitors), antiplatelet medication (eg, clopidogrel), and/or aspirin within 30 days prior to Day 1.
* Subjects with any history of major bleeding or major surgical procedure of any type within 6 months before Day 1.
* Subjects with any history of peptic ulcer, gastrointestinal bleeding including haematemesis, melena, or bleeding from haemorrhoids.
* Subjects with a history of minor bleeding episodes such as epistaxis, rectal bleeding (spots of blood on toilet paper), or gingival bleeding within 3 months before Day 1.
* Subjects who have any family history, suspected or documented, of coagulopathy or haemoglobinopathy or evidence of abnormal coagulation parameters (eg, Prothrombin Time PT, International Normalised Ratio INR or Activated Partial Thromboplastin Time aPTT) at Screening. Subjects with borderline values for PT, INR or aPTT can be enrolled if the abnormality is considered not clinically significant by the investigator.
* Subjects with an estimated glomerular filtration rate (eGFR) at Screening using the MDRD (Modification of Diet in Renal Disease) equation < 90 mL/min.
* Likely possibility that the subject will not cooperate with the requirements of the protocol.
* Objection by General Practitioner to subjects entering the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of DS-1040 | Day 1 to Day 6
  Plasma concentrations of DS-1040 and derived PK parameters up to 6 days after a single 20 mg intravenous infusion of DS-1040.
Cmax Concentration Maximum | Day 1 to Day 6
  derived PK parameters up to 6 days after a single 20 mg intravenous infusion of DS-1040
Tmax time of maximum concentration | Day 1 to Day 6
  derived PK parameters up to 6 days after a single 20 mg intravenous infusion of DS-1040
AUC Area under curve | Day 1 to Day 6
  derived PK parameters up to 6 days after a single 20 mg intravenous infusion of DS-1040
C12h concentration in plasma 12 hours after infusion | Day 1 to Day 6
  derived PK parameters up to 6 days after a single 20 mg intravenous infusion of DS-1040

SECONDARY OUTCOMES:
number and severity of adverse events | Day 1 to Day 6
  safety and tolerability
number and severity of changes in clinical laboratory findings | Day 1 to Day 6
  safety and tolerability
number and severity of changes in physical exam findings | Day 1 to Day 6
  safety and tolerability
number and severity of changes in vital sign findings | Day 1 to Day 6
  safety and tolerability
number and severity of changes in 12-lead electrocardiogram ECG findings | Day 1 to Day 6
  safety and tolerability
change from baseline in thrombin activatable fibrinolysis inhibitor activity | Day 0 (baseline) to Day 6
  Change in baseline of pharmacodynamic parameters (thrombin activatable fibrinolysis inhibitor activity, clot lysis, plasma D-dimer) up to 6 days post dose.tolerability
change from baseline in clot lysis | Day 0 (baseline) to Day 6
  Change in baseline of pharmacodynamic parameters (thrombin activatable fibrinolysis inhibitor activity, clot lysis, plasma D-dimer) up to 6 days post dose.tolerability
change from baseline in plasma D-dimer | Day 0 (baseline) to Day 6
  Change in baseline of pharmacodynamic parameters (thrombin activatable fibrinolysis inhibitor activity, clot lysis, plasma D-dimer) up to 6 days post dose.tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/